CLINICAL TRIAL: NCT03269266
Title: A Multicentre Observational Study to Describe the Prevalence of Scrub Typhus Defined as a Positive Rapid Diagnostic Test Among Selected Patients Presenting With Fever to Clinics in Myanmar
Brief Title: Scrub Typhus RDT Study
Status: Completed | Type: Observational
Sponsor: Myanmar Oxford Clinical Research Unit (Other)
Collaborators: University of Oxford (Other); Medical Action Myanmar (Other); Yae Township Hospital, Mon State (Unknown); Swiss Tropical & Public Health Institute (Other); Defence Services Medical Academy (DSMA), Myanmar (Unknown)
Responsible Party: Sponsor
Other Study IDs: OXTREC 18-17
Record Dates: First submitted 2017-08-29; First posted 2017-08-31 (Actual); Last update posted 2020-01-13 (Actual); Status verified 2019-01

CONDITIONS: The Prevalence of Scrub Typhus
Keywords: Scrub Typhus; Positive Rapid Diagnostic Test
MeSH Terms: conditions — Scrub Typhus

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: Scrub Typhus RDT Test — A transfer pipette or loop will be used to transfer 10 µL of whole blood from a finger prick to the sample pad area on the scrub typhus test strip and the test will be performed on site according to the manufacturer's instructions. Tests will be read by two independent readers and results recorded as positive, negative or invalid.
  In patients with a skin eschar a sterile surgical blade will be used to gently scrape the surface of the eschar. Scrapings will be stored in a cryotube containing 95% ethanol and stored at -80°C for future analysis (PCR genotyping ± whole genome sequencing) to confirm the presence of Orientia tsutsugamushi.

SUMMARY:
Fever is one of most common presenting complaints in clinics in tropical countries. Rickettsial infections, enteric fever and leptospirosis are common and important causes of undifferentiated fever in Southeast Asia. Scrub typhus is caused by Orientia tsutsugamushi and humans are typically infected by a bite of an infected chigger (trombiculid mite larva). Clinical diagnosis is unreliable for identifying scrub typhus, unless a tick eschar is present which is almost pathognomonic for the disease in Southeast Asia. A combination of culture, paired serology and PCR has been proposed as the gold-standard method for detection. As a result laboratory confirmation is not widely available and the diagnosis is missed frequently in clinical practice. Some progress has been made in developing such a test and one promising candidate is the Scrub Typhus Detect IgM Rapid Test (InBios International Inc). We plan to use to this test in this study to estimate the prevalence of scrub typhus in selected febrile patients presenting to clinics in Myanmar .

Patients will be followed up for one week to check for resolution of symptoms.

DETAILED DESCRIPTION:
Title: A multicenter observational study to describe the prevalence of scrub typhus defined as s positive rapid diagnostic test among selected patients presenting with fever to clinics in Myanmar.

Rational and objectives of the study Fever is one of most common presenting complaints in clinics in tropical countries. Rickettsial infections, enteric fever and leptospirosis are common and important causes of undifferentiated fever in Southeast Asia. The largest and earliest reports of scrub typhus in Myanmar were made during World War II when this disease afflicted numerous troops, particularly those serving close to the border with India. Scrub typhus is caused by Orientia tsutsugamushi and humans are typically infected by a bite of an infected chigger (trombiculid mite larva). Clinical diagnosis is unreliable for identifying scrub typhus, unless a tick eschar is present which is almost pathognomonic for the disease in Southeast Asia. A combination of culture, paired serology and PCR has been proposed as the gold-standard method for detection. As a result laboratory confirmation is not widely available and the diagnosis is missed frequently in clinical practice. Some progress has been made in developing such a test and one promising candidate is the Scrub Typhus Detect IgM Rapid Test (InBios International Inc). In laboratory-based evaluations using stored sera collected from patients recruited in a study in Thailand with confirmed scrub typhus this test had a sensitivity of ~80% for the detection of the disease compared to serological methods. We plan to use to this test in this study to estimate the prevalence of scrub typhus in selected febrile patients presenting to clinics in Myanmar.

Primary objective: To describe the prevalence of scrub typhus defined as a positive rapid diagnostic test among selected patients presenting with fever to clinics in Myanmar

Secondary objective:

* To assess inter-observer agreement when interpreting the tests
* To assess the ease-of-use of the tests
* To direct future research efforts into rickettsial disease in Myanmar
* To raise awareness of the presence of scrub typhus in Myanmar Inclusion criteria

  1. Male or female >1 year of age
  2. Fever defined as > 38 °C tympanic temperature
  3. Duration of fever >48h
  4. Written informed consent (by legally acceptable representative in case of children), and assent for children age 10-17 year
  5. Eschar (60 patients only) Exclusion criteria
* Malaria confirmed by RTD or microscopy
* Skin/soft tissue infection, dysentery or urinary tract infection probable cause of fever

Procedures and Methodology The study will be carried out to describe the prevalence of scrub typhus defined as a positive rapid diagnostic test among patients presenting with fever to six participating clinics in Myanmar.

Patients coming with fever to participating clinics will be routinely assessment by attending physician. Patients meeting the inclusion and exclusion criteria for the study will be invited and enrolled to the study after getting informed consent.

Rapid diagnostic test and laboratory procedure A scrub typhus rapid test will be performed on site by using the InBios Scrub Typhus Detect IgM Rapid Test. Tests will be read by two independent readers and results recorded as positive, negative or invalid. In case of invalid test result, another test will be performed using a new test strip. If there is any disagreement between two readers, the lead investigator at the site will decide the test result and the test will be photographed.

In patients with a skin eschar a sterile surgical blade will be used to gently scrape the surface of the eschar. Scrapings will be stored in a cryotube containing 95% ethanol and stored at -80°C for future analysis (PCR genotyping ± whole genome sequencing) to confirm the presence of Orientia tsutsugamushi.

Treatment Physicians will be advised to formulate a treatment plan according to their usual practice but it will be recommended that treatment for scrub typhus be added to the regimen if the test is positive i.e. doxycycline 100mg bd for seven days in adults or 4mg/kg day in two divided doses in children older than eight years. Doxycycline is contraindicated in pregnant women and children eight years old or below and these groups should be prescribed azithromycin (500mg single dose).

Follow up Patients will be reassessed at one week to check for resolution of fever and symptoms . Any patient with ongoing symptoms will be re-assessed by a physician.

Duration and Study Sites Patients will be recruited 1 year starting from December 2017 to November 2018 in six sites: Yae township hospital, No.2, 1000 Bedded Military Hospital (Nay Pyi Taw), No.20, 100 Bedded Military Hospital (Tha Beik Kyin), NAP-MAM clinics (Kawkareik and Putao township), No.2, 300 Bedded Military Hospital (Ann, Rakhine State).

Risk and benefits This is a low risk study. Finger prick for RDT and scrapping from eschar (for patients who have eschar) may cause slight discomfort. Some patients may receive antibiotics they would not have otherwise been prescribed as a result of having the test. However this is most likely to benefit them as these tests have been shown to be sensitive and specific for the diagnosis of scrub typhus in similar settings.

Incentives and Compensation There will be no incentives or compensation for study participation. Confidentiality The study will ensure that the participants' anonymity is maintained. The participants will be identified only by initials and a study number on the CRF and the study database.

Publication The research findings will be disseminated to policy-makers and other interested parties inside Myanmar. If there are any publications resulting from the results all those who have made a substantial contribution will be co-authors.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female >1 year of age
2. Fever defined as > 38 °C tympanic temperature
3. Duration of fever (self-reported) >48h
4. Written informed consent (by parent or legally acceptable representative in case of children), and assent for children aged 10-17 years
5. Eschar (60 patients only)

Exclusion Criteria:

1. Malaria confirmed by RDT or microscopy
2. Skin/soft tissue infection, dysentery or urinary tract infection probable cause of fever

Min Age: 1 Year | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients with fever (± eschar) presenting to community health clinics/hospitals in Myanmar
Sampling Method: Probability Sample
Enrollment: 136 (Actual)
Dates: Start 2017-12-04 (Actual); Primary Completion 2019-12-26 (Actual); Study Completion 2019-12-26 (Actual)

PRIMARY OUTCOMES:
Positive RDT Result | 15 Minutes
  Proportion of patients with a positive RDT result

SECONDARY OUTCOMES:
Inter-observer agreement expressed as the kappa statistic | 15 Minutes
  Ease- of- use of the test (scored on blood safety, quality of instructions, number of timed steps to perform test, ease of interpretation, user satisfaction)
Fever/symptom resolution | One Week
  Proportion of patients with fever/symptom resolution at one week

CONTACTS AND LOCATIONS:
Overall Officials: Elizabeth Anne Ashley, Dr, Study Director — Myanmar Oxford Clinical Research Unit; Ni Ni Tun, Dr, Study Director — Medical Action Myanmar; Aye Thida Aye, Dr, Study Director — Yae Township Hospital, Mon State; Kyaw Myo Tun, Dr, Study Director — Defence Services Medical Academy (DSMA); Khine Khine Su, Prof, Study Director — Defence Services Medical Academy (DSMA); James Heaton, Dr, Study Director — Myanmar Oxford Clinical Research Unit; Kyaw Soe, Study Director — Myanmar Oxford Clinical Research Unit; Daniel Paris, Prof, Study Director — Swiss Tropical & Public Health Institute; Frank Smithuis, Prof, Principal Investigator — Myanmar Oxford Clinical Research Unit and Medical Action Myanmar; Myo Mg Mg Swe, Dr, Study Director — Myanmar Oxford Clinical Research Unit
Locations (2):
- Burma (2):
  - No.20, 100 Bedded Military Hospital,, Thabeikkyin, Mandalay Region
  - No.2, 1000 Bedded Military Hospital, Nay Pyi Taw